CLINICAL TRIAL: NCT02655484
Title: Evaluation of Carbon Dioxide Rebreathing During Exercise Assisted by Non-invasive Ventilation
Brief Title: Carbon Dioxide Rebreathing During Exercise Assisted by Non-invasive Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, RongChang Chen, director of Guangzhou Institute of Respiratory Disease, Guangzhou Institute of Respiratory Disease
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2009CB522112
Record Dates: First submitted 2016-01-06; First posted 2016-01-14 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; noninvasive ventilation; exercise; CO2 rebreathing
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- COPD patients (Other): Oxygen was delivered to the face mask by a tube at a constant rate (5L/min) to keep the fingertip oxygen saturation at 90% or above. Ventilatory assistance was delivered using a BiPAP® Vision® ventilator (Respironics, Murrysville, Pennsylvania, USA) in BiPAP mode applied via a tightly fitting full face mask (Curative, Suzhou, China). A symptom-limited cycle exercise test was performed while assisted by non-invasive ventilation (NIV). All measurements were recorded at inspiratory pressure of 14 cmH2O, expiratory pressure of 4 cmH2O during rest and exercise. Breathing pattern, mean exhalation flow, mean plateau exhalation valve flow, the mean inspiratory fraction of CO2 (tidal FiCO2) reinsufflated from the circuit between the mask and the exhalation valve was measured for each breath.
  Interventions: Device: BiPAP® Vision® ventilator（"Ventilator", "Philips Respironics™ BiPAP® Vision®" ）

INTERVENTIONS:
Device: BiPAP® Vision® ventilator（"Ventilator", "Philips Respironics™ BiPAP® Vision®" ） — See details from arm descriptions.

SUMMARY:
The purpose of this study was to evaluate whether CO2 rebreathing occurs in healthy subjects or patients with COPD ventilated during exercise assisted by the single-limb circuit with a plateau exhalation valve at a given inspiratory positive airway pressure and a minimal level of expiratory positive airway pressure (EPAP) and whether there is a potential threshold for predicting CO2 rebreathing.

DETAILED DESCRIPTION:
Non-invasive ventilation circuit consists of single-limb tubing for inspiration and expiration, including a plateau exhalation valve. As exhaled gases was vented out the plateau exhalation valve at a constant rate, during exercise, with the increase of exhalation flow, single-limb circuit with a plateau exhalation valve might cause carbon dioxide(CO2) rebreathing. Therefore, our aim in the present study was to evaluate whether CO2 rebreathing occurs in COPD patients ventilated during exercise assisted by the single-limb circuit with a plateau exhalation valve and estimate a potential threshold for predicting CO2 rebreathing.

ELIGIBILITY:
Inclusion Criteria:

* presented clinically stable (no exacerbation in the 4 weeks prior to study participation or with no change in medications);
* physician diagnosed COPD, forced expiratory volume in 1s (FEV1) < 50% predicted;
* dyspnea as a main symptom that limited daily activities.

Exclusion Criteria:

* subjects with obvious pulmonary bullae demonstrated by chest CT scan or X-ray;
* examination or facial trauma/malformation, recent facial, upper airway or upper gastrointestinal tract surgery, that would preclude receiving NIV therapy;
* a history of coronary artery disease or cardiac arrhythmias or potential electrocardiographic alterations;
* a history of uncontrolled hypertension, or other respiratory diseases;
* oxygen saturation(SpO2) < 88% at rest with a fraction of inspired oxygen (FiO2) ≥ 0.5;
* patients with musculoskeletal or neurological disorders;
* or failure to comply with the research protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
mean exhalation valve flow | Measurements were collected continuously throughout a symptom-limited cycle exercise test （test lasts for about 8-12 min） while subjects breathed through the full face mask. Analyses were made breath by breath during the whole test process.

SECONDARY OUTCOMES:
mean exhalation flow | Measurements were collected continuously throughout a symptom-limited cycle exercise test （test lasts for about 8-12 min） while subjects breathed through the full face mask. Analyses were made breath by breath during the whole test process.
mean inspiratory fraction of CO2 for each tidal volume | Measurements were collected continuously throughout a symptom-limited cycle exercise test （test lasts for about 8-12 min） while subjects breathed through the full face mask. Analyses were made breath by breath during the whole test process.
fraction of end-tidal carbon dioxide partial pressure | Measurements were collected continuously throughout a symptom-limited cycle exercise test （test lasts for about 8-12 min） while subjects breathed through the full face mask. Analyses were made breath by breath during the whole test process.
inspiratory time | Measurements were collected continuously throughout a symptom-limited cycle exercise test （test lasts for about 8-12 min） while subjects breathed through the full face mask. Analyses were made breath by breath during the whole test process.
expiratory time | Measurements were collected continuously throughout a symptom-limited cycle exercise test （test lasts for about 8-12 min） while subjects breathed through the full face mask. Analyses were made breath by breath during the whole test process.
respiratory rate | Measurements were collected continuously throughout a symptom-limited cycle exercise test （test lasts for about 8-12 min） while subjects breathed through the full face mask. Analyses were made breath by breath during the whole test process.
inspiratory tidal volume | Measurements were collected continuously throughout a symptom-limited cycle exercise test （test lasts for about 8-12 min） while subjects breathed through the full face mask. Analyses were made breath by breath during the whole test process.
expiratory tidal volume | Measurements were collected continuously throughout a symptom-limited cycle exercise test （test lasts for about 8-12 min） while subjects breathed through the full face mask. Analyses were made breath by breath during the whole test process.

CONTACTS AND LOCATIONS:
Overall Officials: Rongchang Chen, MD, Principal Investigator — Guangzhou Institute of Respiratory Disease
Locations (1):
- State Key Laboratory of Respiratory Disease, First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China